CLINICAL TRIAL: NCT07178691
Title: A Precision Medicine Approach to the Prevention of Depression in Patients With Atrial Fibrillation - HOPE-AF
Brief Title: A Precision Medicine Approach to the Prevention of Depression in Patients With Atrial Fibrillation
Acronym: HOPE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Aalborg University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12.048; S-20230078 (Other: Committees on Health Research Ethics for Southern DK (VEK))
Record Dates: First submitted 2025-08-26; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF); Depression - Major Depressive Disorder; Anxiety
Keywords: atrial fibrillation; prevention of depression; Psychological intervention; online intervention
MeSH Terms: conditions — Atrial Fibrillation; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- online psychological intervention (Experimental): The participants will receive the HOPE-AF online psychological intervention. The intervention is designed to prevent depression in patients with atrial fibrillation
  Interventions: Other: Online psychological intervention

INTERVENTIONS:
Other: Online psychological intervention — The HOPE-AF intervention is an online psychological intervention to prevent depression in patients with atrial fibrillation. The intervention combines verbal psychological sessions over phone or video with online text messages and a tailored 4-12 weeks online intervention with new modules each week including psychological exercises in writing and as sound exercises (e.g., breathing exercises and relaxations exercises etc.) and videos.

SUMMARY:
The purpose of the proposed project is to test a new therapist-assisted, eHealth intervention (HOPE-AF) targeted to prevent depression in patients with atrial fibrillation (AF). AF is the most common sustained cardiac arrhythmia. Age is the most common risk factor for AF, and given the ageing of the population, the prevalence of AF has increased threefold during the last 50 years. AF is now considered a major public health challenge. AF is not only associated with increased risk of stroke and heart failure but patients with AF also tend to continuously focus on the body's signals and have difficulties accepting the disease. This is often paired with psychological reactions, such as excessive worry and anxiety, increasing the risk of withdrawal from social activities, which often leads to depression. Patients with AF and comorbid depression are at greater risk of a poor prognosis.

The project is a feasibility study to examine acceptability, adherence and limited efficacy, as well as barriers and facilitators for implementation of the intervention in clinical practice. The project is multi-disciplinary and embedded within the rehabilitation setting in the hospitals, enhancing the chance of later implementation.

DETAILED DESCRIPTION:
HOPE-AF represents a novel and pioneering approach to improving the HRQoL and prognosis of patients with AF through the prevention of depression, a seminal and debilitating risk factor for the onset of AF and worsening AF prognosis. Together with patients, the investigators co-designed an online psychological intervention that targets risk factors for depression with respect to preventing depression.

The feasibility of the intervention in clinical practice will be assessed. The intervention will be delivered via a GDPR-secured platform. This is an innovative solution for care delivery, enabling patients to access the intervention anytime, which may enhance adherence due to the flexibility of access and delivery. The investigators has previously shown that this eHealth mode of delivery is well received by patients.

Meta-analyses show that online psychological interventions are effective in preventing depression and anxiety in both at-risk cohorts and the general population. These positive effects have been shown for the cognitive-behavioral, interpersonal, and positive psychology therapeutic approaches.

The HOPE-AF intervention Recent research demonstrates that personalizing the prevention of depression by targeting individual risk factors for the disorder in every single patient can optimize treatment outcomes. HOPE-AF will specifically target and remediate the core risk factors for depression of each enrolled individual patient (i.e., stress, loneliness, social isolation, anhedonia, lack of exercise, low self-esteem, rumination, anxiety and sleep problems), using existing evidence-based treatments and a precision medicine approach to prevent depression.

The intervention is co-developed with patients and health professional and targeted to AF patients without current depression and anxiety. The intervention modules consist of psychoeducation, psychological tools, psychological therapies targeted to patients' risk factors for depression, and multimedia contents and exercises. Patients will complete the modules online and be assisted by a therapist who will provide feedback through asynchronous text messages via a GDPR secured platform. Phone or video (according to patients´ preferences) consultations with the therapist as add-on to the online intervention will be possible on a need to basis. The treatment duration will vary from patient to patient depending on the prevalent risk factors for depression and the severity of the risk factors. The duration will range from 4-12 weeks, as some modules will be mandatory for all patients, while other modules will only be relevant to target specific risk factors. Patients are expected to spend 1-2 hours per week on a module.

The HOPE-AF intervention is based on several different forms of evidence-based psychotherapies, including Cognitive Behavioral Therapy (CBT), Metacognitive Therapy (MCT), Acceptance and Commitment Therapy (ACT), Compassion Focused Therapy (CFT), Existential Therapy, Mindfulness, Interpersonal Therapy (IPT) and YOGA with psychological components. The included therapies allow for the most effective and comprehensive way of "treating" each specific risk factor for depression in each individual patient, with respect to patients' needs and preferences. Therapists also administer the CORE-10 questionnaire to patients every week during the intervention to evaluate progress. In case of deterioration, a contingency plan as written into the treatment protocol will be implemented that includes e.g., more frequent contact, more tailoring to meet patients' needs, suicidal risk assessment, and if relevant referral to the patient's GP. If patients become ill or leave on holidays during the intervention, the duration of the intervention will be extended with up to three weeks.

OBJECTIVES AND HYPOTHESES The overall purpose of HOPE-AF is to prevent depression and improve the health outcomes of patients with AF.

Specific objectives of the HOPE-AF feasibility study are to:

* Assess the feasibility of the HOPE-AF intervention, with respect to acceptability and adherence, limited efficacy and patient retention (barriers and facilitators).
* To test procedures with respect to recruitment and implementation in clinical practice.

INCLUSION Eligible patients will be included from cardiac units at hospitals. Patients are screened for symptoms of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS) questionnaire (range 0-21 for depression and anxiety respectively with increasing score reflecting more symptoms). Patients with HADS-D ≥11 or HADS-A ≥11, [which is considered a clinically significant level of symptoms] will be excluded from the study, since this a prevention initiative and not treatment. Eligible patients will receive the baseline questionnaire. Patients who do not complete the questionnaire within 30 days, will be excluded.

After completion of the baseline questionnaire, patients will be subjected to a brief standardized telephone interview by a member of the HOPE-AF team to further check for eligibility. The interview will be used to confirm patients´ motivation for participation, assess if patients have reading/writing abilities and internet literacy enabling adherence to the intervention, assess if patients are able to spend 1-2 hours on the intervention each week, and to assess if other life circumstances (e.g., present somatic health problems or other stressors in their personal life) make it impossible to adhere sufficiently to the intervention, and to exclude patients with a need for psychiatric help due to comprehensive psychiatric issues or major psychopathology. If patients answer yes to at least 1 of 3 purpose-designed questions to screen for suicidal ideation in the baseline questionnaire, the psychologist will make further assessments to determine if the patient requires psychiatric treatment.

To determine present risk factors for depression, eligible patients will receive a diagnostic interview by their assigned therapist. The presence or absence of risk factors for depression will determine the length and content of the HOPE-AF intervention.

DATA Given the general purpose of the feasibility study to examine barriers and facilitators related to the intervention and later successful implementation, the investigators will primarily use descriptive statistics (e.g., frequencies, percentages, means, ranges, and standard deviations) to analyse the patients pre-post outcome data and to estimate recruitment and data retention rate. The collected outcome measures are described elsewhere.

The feasibility study will also include interviews post-intervention with a sample of 10 participants, using semi-structured interviews related to their experiences with the intervention and procedures. The interview guide includes questions related to patient satisfaction, acceptance of the intervention, and barriers and facilitators for later implementation in clinical practice at a patient and organizational level. Interviews will be transcribed and analyzed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of paroxysmal or persistent AF [if persistent AF, duration < 2 years]
* Able to use and access a computer or tablet/iPad to adhere to the intervention - Proficient in the Danish language (reading and writing)
* Ability to provide informed written consent.

Exclusion Criteria:

* Depression [Hospital Anxiety and Depression Scale: HADS-D ≥11 (moderate symptoms)
* Anxiety [Hospital Anxiety and Depression Scale: HADS-A ≥11 (moderate symptoms)
* Severe psychiatric or neurological disorder (e.g., schizophrenia or dementia)
* In need of psychiatric help due to comprehensive psychiatric issues, diagnosed or not
* Seeing a psychologist or mental health professional for the treatment of depression and anxiety
* Experiencing significant life stressors that hinder adherence to the HOPE-AF treatment
* Participating in another research project involving intervention for depression
* Not being able or willing to spend 1-2 hours on the intervention each week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Drop out rate | From start of the intervention to completion of intervention, i.e., from 0 to 12 weeks.
  Drop out rate. What is the rate of drop out during the intervention from the 28 included patients. Drop out is defined as patients who want to stop the intervention or patients who stop responding to messages and phone/video calls. A drop-out rate <25% was considered acceptable.

SECONDARY OUTCOMES:
Adherence | From start of the intervention to completion of intervention, i.e., from 0 to 12 weeks.
  The rate of completion of the assigned modules. Each module was labelled completed or non-completed. Completion of each module was defined as having completed tasks in the module and communicated with the therapist about the content.
Symptoms of depression | From completion of baseline questionnaire (after enrollment and prior to intervention start) to completion of follow up questionniare (sent to patients 13 weeks after intervention start).
  Mean change score from baseline to follow-up on Depression (Hospital Anxiety and Depression Scale) (HADS-D). Range from 0-21 with higher score indicating more symptoms.
Anxiety related to cardiac disease | From completion of baseline questionnaire (after enrollment and prior to intervention start) to completion of follow up questionniare (sent to patients 13 weeks after intervention start).
  Mean change score of Anxiety related to cardiac disease (Cardiac Anxiety Questionnaire (CAQ)) from baseline to follow-up.
  CAQ comprises 18 items and can be divided in three subscales (Fear, 8 items; Avoidance, 5 items; Attention, 5 items). Each item is scored from 0 (never) to 4 (always). Higher score indicates greater number of symptoms or greater frequency. The total score is divided by the number of items, making the score range from 0 to 4 for each subscale and the total score.
Symptoms of anxiety | From completion of baseline questionnaire (after enrollment and prior to intervention start) to completion of follow up questionniare (sent to patients 13 weeks after intervention start).
  Mean change score of Anxiety from baseline to follow-up:
  Anxiety (Hospital Anxiety and Depression Scale) (HADS-A). Range from 0-21 with higher score indicating more symptoms.
Atrial fibrillation related quality of life | From completion of baseline questionnaire (after enrollment and prior to intervention start) to completion of follow up questionniare (sent to patients 13 weeks after intervention start).
  Mean change score from baseline to follow-up on: Atrial Fibrillation Effect on QualiTy-of-life Questionnaire (AFEQT) including total score and subscales (symptoms, daily activities, treatment concern). Total score and subscales range from 0-100 with higher score indicating better score.
AF symptom burden | From completion of baseline questionnaire (after enrollment and prior to intervention start) to completion of follow up questionniare (sent to patients 13 weeks after intervention start).
  Mean change score from baseline to follow-up on: AF symptom burden (AF-6). Range from 0-60 with higher score indicating worse outcome.
Health related Quality of Life | From completion of baseline questionnaire (after enrollment and prior to intervention start) to completion of follow up questionniare (sent to patients 13 weeks after intervention start).
  Mean change score from baseline to follow-up on: Health related Quality of Life (HeartQoL quesionnaire). The HeartQoL questionnaire is a 14-item questionnaire consisting of a Global scale [14 items] made up of Physical [10 items] and Emotional [4 items] subscales. Each subscore ranges from 0-3, a higher score indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne s Pedersen, Professor, Principal Investigator — University of Southern Denmark, Department of Psychology
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - University Hospital Esbjerg and Grindsted, University of Southern Denmark, Esbjerg
  - Zealand University Hospital, Roskilde, Department of Cardiology, Roskilde

IPD SHARING:
Plan to Share IPD: No